CLINICAL TRIAL: NCT04162613
Title: Sensorimotor Function as Predictor for Graft Rupture After Anterior Cruciate Ligament Reconstruction: A Prospective Cohort Study (STOP Graft Rupture)
Brief Title: Can Sensorimotor Function Predict Graft Rupture After ACL Reconstruction
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: STOP Graft Rupture
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior cruciate ligament injury; re-injury; muscle function; functional performance; rehabilitation; physiotherapy; sensorimotor control
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Reinjuries | interventions — Muscle Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ACL reconstruction in Lund and Umeå: Persons who have suffered a unilateral anterior cruciate ligament injury treated with reconstruction
  Interventions: Other: Different measures of muscle function such as muscle strength, hop tests, postural orientation and muscle activation

INTERVENTIONS:
Other: Different measures of muscle function such as muscle strength, hop tests, postural orientation and muscle activation — The participants will be assessed with a physical test battery at baseline including: Isokinetic knee strength, Isometric strength of trunk and lower extremity, Single-leg hop for distance, side hop, postural orientation (single leg-squat, stair descending, forward lunge, Single-leg hop for distance, side-hop), hip and ankle range of joint motion, muscular activation pattern, 3D movement analysis and proprioception test.
  At follow-up (2 years), the participants will be asked to answer a survey about new ACL injuries and return to sport/previous activity level.

SUMMARY:
In this longitudinal prospective cohort study including young people with anterior cruciate ligament (ACL) reconstruction, the investigators will evaluate if poor sensorimotor function at baseline can predict 1) graft rupture 2) the risk of contra-lateral ACL injury and 3) failure to return to sport/previous activity level within 3 years following ACL reconstruction.

DETAILED DESCRIPTION:
In this longitudinal prospective cohort study including young athletic men and women (aged 15-35) with ACL reconstruction (ACLR), it will be investigated if poor sensorimotor function at baseline (1 year post ACLR), such as hop performance, muscle strength and postural orientation can predict 1) graft rupture 2) the risk of contra-lateral ACL injury and 3) failure to return to sport/previous activity level within 3 years following ACLR.

Statistics Separate logistic regression models will be used to elucidate the influence of each muscle sensorimotor function variable on the outcomes (graft rupture, contra-lateral injury, return to sport/activity level failure), adjusted for potential confounders. With the LSI for the single-leg hop test as main outcome, power calculations show that with a re-injury rate of 7%, an estimated odds ratio of 0.95, power=80% and alpha=5 %, at least 174 individuals are needed. Based on this calculation, 200 individuals will be included for the prospective analysis, allowing for an approximate drop-out of 10%.

ELIGIBILITY:
Inclusion Criteria:

* 8-16 months after ACL reconstruction
* With or without associated injuries to other structures of the knee (e.g., collateral ligament(s), meniscal injury)
* Age 15-35 years.

Exclusion Criteria:

* ACL injury other knee and previous ACL injury index knee
* Diseases or disorders overriding the knee condition (e.g., neurological or rheumatological disease)
* Not understanding the languages of interest (any Scandinavian language or English).

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be recruited from the Department of Orthopedics, Norrland University hospital, Umeå, Sweden and Skåne University Hospital, Lund, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with graft rupture | 2 years
  Number of patients that have sustained a rupture of the reconstructed ligament

SECONDARY OUTCOMES:
Number of patients with contra-lateral ACL injury | 2 years
  Number of patients that have sustained an injur to the contra-lateral knee
Failure to return to sport/previous activity level | 2 years
  Number of patients that had failed to return to previous sport/activity level

CONTACTS AND LOCATIONS:
Overall Officials: Anna Cronström, PhD, Principal Investigator — Umeå University; Charlotte Häger, Professor, Study Chair — Umeå University
Locations (1):
- UMotion laboratory, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cronstrom A, Ageberg E, Hager CK. Does sensorimotor function predict graft rupture, contra-lateral injury or failure to return to sports after ACL reconstruction? A protocol for the STOP Graft Rupture study. BMJ Open. 2021 Jan 8;11(1):e042031. doi: 10.1136/bmjopen-2020-042031. PMID 33419913